CLINICAL TRIAL: NCT01315990
Title: Non-randomized Phase-IV-study to Investigate the Efficacy of FOLFIRI in Combination With Cetuximab in the First-line Treatment of Metastatic Colorectal Cancer Including a Regular Dermal Prophylaxis to Prevent Acneiforme Follicular Exanthema
Brief Title: FOLFIRI in Combination With Cetuximab in the First-line Treatment of Metastatic Colorectal Cancer Including a Regular Dermal Prophylaxis to Prevent Acneiforme Follicular Exanthema
Acronym: DERMATUX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Carl Schimanski (Other)
Responsible Party: Sponsor-Investigator, Dr. Carl Schimanski, Principal Investigator, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DERMATUX
Record Dates: First submitted 2011-03-11; First posted 2011-03-16 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Phase IV Study; Metastatic Colorectal Cancer (mCRC; Cetuximab (Erbitux); first-line treatment; acneiform follicular exanthema; rash; vitamin K1
MeSH Terms: conditions — Colorectal Neoplasms; Exanthema | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRI + Cetuximab (Experimental)
  Interventions: Drug: FOLFIRI + Cetuximab

INTERVENTIONS:
Drug: FOLFIRI + Cetuximab — 1. Cetuximab (Erbitux® )- Cetuximab is a recombinant IgG1 chimeric monoclonal antibody directed against human epidermal growth factor receptor (EGFR).
  2. FOLFIRI regimen
  Administration Schedule:
  Cetuximab at a initial dose 400 mg/sqm (first week), then 250 mg/sqm on day 1 and 8 Background Chemotherapy (every two weeks)
  * Irinotecan 180 mg/m² iv , 90 min on day 1
  * Folic acid (racemic) 400 mg/m², 120 min on day 1
  * 5-FU 400 mg/m² bolus on day 1
  * 5-FU 2400 mg/m² iv over 46 h on day 1 to 2

SUMMARY:
The purpose of this interventional study is to assess the progression free survival (one year) of patients with treatment of FOLFIRI and cetuximab, combined with an optional dermal prophylaxis.

Further Objectives:

1. Development of acneiforme follicular exanthema >= grade 2
2. Duration until development of acneiforme follicular exanthema >= grade 2
3. Development of paronychia
4. Development skin fissure (hand and foot)
5. Objective remission according RECIST 1.1
6. Rate of secondary resections of liver metastasis with a curative approach
7. Assessment of safety and tolerability
8. Overall survival
9. Progression free survival

DETAILED DESCRIPTION:
Subjects with metastatic colorectal cancer and confirmed KRAS-wildtype status in 1st line therapy will be included in this phase IV-study. Subject will receive a regimen of FOLFIRI in combination with Cetuximab every two weeks during study treatment phase. Treatment continues until

* disease progression
* complete response
* development of status of operability
* an uncontrollable exanthema grade 3 or 4 or
* intolerable toxicity is diagnosed. After study discontinuation or end of treatment, respectively, patients will be followed up until the the last patient was treated for 12 months and has completed the 36-months follow up phase. Tumor response will be evaluated (according to RECIST 1.1) every 12 weeks and at the end of study treatment

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed metastatic colorectal cancer (primary tumor or metastasis)
* Confirmation of KRAS wildtype status
* Confirmation of EGFR-Expression in the tumor
* Stadium IV
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Qualified for an application of FOLFIRI + Cetuximab treatment
* Signed patient informed consent form
* Of either gender and aged 18 years or more
* Estimated lifespan more than 3 months
* Measurable disease according to RECIST 1.1 guidelines. The evaluation has to be max. 4 weeks
* Effective and adequate contraceptive precautions of man or woman in a childbearing potential age (double barrier method)
* Leucocytes ≥ 3,0 x 10^9/L with neutrophils ≥ 1,5 x 10^9/L, thrombocytes ≥ 100 x 10^9/L, haemoglobin ≥ 5,6 mmol/L
* Serum bilirubin ≤ 1,5 x ULN (upper limit of normal)
* ALAT and ASAT ≤ 2,5 x ULN; if metastasis in liver, than ALAT and ASAT ≤ 5 x ULN
* Serum creatinin ≤ 1,5 x ULN
* If applicable a prior operation has to be min. 4 weeks ago, biopsy more than 1 week until initiation of treatment. Wounds of operations had to be completely cured
* No toxicity of prior treatments

Exclusion Criteria:

* KRAS-gene mutation
* Confirmation of non-EGFR-Expression
* Prior treatment with an EGRF-receptor inhibitor
* Prior chemotherapy of the mCRC, except (neo-)adjuvant therapy, which had to be ended min. 6 months before recruitment
* Experimental treatment medication within 30 days before recruitment
* Known hypersensitivity against components of the chemotherapy, cetuximab, doxycycline, Reconval K1 or Dermatop
* Rosacea
* Other chronic dermal diseases with development of papula or pustule
* Known lung fibrosis or interstitial pneumonitis or interstitial lung diseases
* keratitis, ulcerative keratitis or severe form of dry eye
* Pregnancy or breast feeding
* Brain metastasis
* Clinical relevant coronary heart disease, myocardial infarction within the last 12 months or high risk of uncontrollable arrhythmia
* Acute or subacute ileus or chronic colon-inflammation or chronic diarrhea
* Symptomatic peritoneal carcinomatosis
* Serious, non-healing wounds, ulcera or bone fractures
* Uncontrollable arterial hypertension
* Therapeutic anticoagulation (e.g. therapy with marcumar)
* Known dihydropyrimidine dehydrogenase deficiency
* Gilbert-Meulengracht-syndrome
* Other malignant tumours less than five years old. Exceptions include basocellular carcinoma or an in situ cancer of the cervix uteri if they are curative treated as well as an untreated, locally confined, asymptotic "low risk" (indolent) prostata carcinoma (Stage T ≤ T1-2a, PSA < 15 ng/ml, Gleason-Score ≤ 6 ).
* Known abuse of narcotic drugs or alcohol
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with the study procedures
* Any significant concomitant disease that excludes the participation to the study
* Missing or limited juristic contractual capability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 12 months
  Progression-free survival rate at 12 months

SECONDARY OUTCOMES:
Progression-free survival | up to end of follow-up-phase (36 months)
ORR | approximately 12 months
  Objective response rate over the entire treatment period
OS | The time from regsitration date to the date of death
  Overall survival time
Duration until development of acneiforme follicular exanthema >= grade 2 | approximately 12 months
  Duration until development of acneiforme follicular exanthema >= grade 2 during treatment-phase
Development of paronychia | approximately 12 months
  Development of paronychia during treatment-phase
Development of skin fissure (hand and foot) | approximately 12 months
  Development of skin fissure (hand and foot) during treatment-phase
Rate of secondary resections of metastasis of liver with a curative approach | approximately 12 months
  Rate of secondary resections of metastasis of liver with a curative approach during treatment-phase
Assessment of safety and tolerability | approximately 12 months
  Assessment of safety and tolerability during treatment phase
Development of acneiforme follicular exanthema >= grade2 | approximately 12 months
  Development of acneiforme follicular exanthema >= grade2 during treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: Carl Christoph Schimanski, PD Dr. med., Principal Investigator — Universitätsmedizin Mainz
Locations (1):
- Universitätsmedizin Mainz, Mainz, Germany